CLINICAL TRIAL: NCT00435110
Title: Effects of PEEP and FiO2 in the Evaluation of Severity of ALI and ARDS
Brief Title: Effects of PEEP and FIO2 in ALI and ARDS
Acronym: HELP
Status: Completed | Type: Observational
Sponsor: Instituto Canario de Investigacion Biomedica (Other)
Collaborators: Asociación Científica Pulmón y Ventilación Mecánica (Other)
Other Study IDs: 22
Record Dates: First submitted 2007-02-12; First posted 2007-02-14 (Estimated); Last update posted 2018-10-11 (Actual); Status verified 2018-10

CONDITIONS: Acute Respiratory Distress Syndrome; Acute Lung Injury; Acute Respiratory Failure
Keywords: ARDS; ALI; Mechanical Ventilation; Outcome
MeSH Terms: conditions — Respiratory Distress Syndrome; Acute Lung Injury | interventions — Positive-Pressure Respiration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

INTERVENTIONS:
Procedure: standard ventilatory settings
Procedure: PEEP and FiO2

SUMMARY:
Current American-European Consensus Conference (AECC) definitions for ALI and ARDS are inadequate for inclusion into clinical trials due to the lack of standardization for measuring the oxygenation defect. We questioned whether an early assessment of oxygenation on specific ventilator settings would identify patients with established ARDS (persisting over 24h).

DETAILED DESCRIPTION:
We designed this study to determine whether standard ventilator settings applied on the day ARDS is identified (Day 0) or 24 hours (Day 1) later: (1) would have an impact on the reclassification of patients into ALI or ARDS, and (2) would identify groups with different clinical outcomes. Our hypothesis was that the assessment of PaO2/FiO2 on standard ventilator settings 24 hours after patients originally met the AECC definition of ARDS would identify patients with established ARDS (persisting over 24 h) from others with different degrees of lung injury. If this hypothesis is supported, it would suggest that patients with a better outcome could have been preferentially entered into one group of previously conducted clinical trials, resulting in a viable therapy being proved useless or useless therapy proven viable.

ELIGIBILITY:
Inclusion Criteria:

* All patients meeting American-European Consensus Conference (AECC) ARDS criteria were approached for enrollment regardless of their current status or past medical history.

Exclusion Criteria:

* The only patients excluded were those in which >24 hrs had pasted after initially meeting the AECC ARDS criteria before consent and results of initial standard ventilator settings could be obtained.

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 178 (Actual)
Dates: Start 2004-05; Study Completion 2005-10

CONTACTS AND LOCATIONS:
Overall Officials: Jesus Villar, MD, PhD, Principal Investigator — Instituto Canario de Investigación Biomédica
Locations (1):
- Hospital Universitario NS de Candelaria, Santa Cruz de Tenerife, Canary Islands, Spain

REFERENCES:
- [Derived] Villar J, Ambros A, Mosteiro F, Martinez D, Fernandez L, Ferrando C, Carriedo D, Soler JA, Parrilla D, Hernandez M, Andaluz-Ojeda D, Anon JM, Vidal A, Gonzalez-Higueras E, Martin-Rodriguez C, Diaz-Lamas AM, Blanco J, Belda J, Diaz-Dominguez FJ, Rico-Feijoo J, Martin-Delgado C, Romera MA, Gonzalez-Martin JM, Fernandez RL, Kacmarek RM; Spanish Initiative for Epidemiology, Stratification and Therapies of ARDS (SIESTA) Network. A Prognostic Enrichment Strategy for Selection of Patients With Acute Respiratory Distress Syndrome in Clinical Trials. Crit Care Med. 2019 Mar;47(3):377-385. doi: 10.1097/CCM.0000000000003624. PMID 30624279
- [Derived] Villar J, Martinez D, Mosteiro F, Ambros A, Anon JM, Ferrando C, Soler JA, Montiel R, Vidal A, Conesa-Cayuela LA, Blanco J, Arrojo R, Solano R, Capilla L, Del Campo R, Civantos B, Fernandez MM, Aldecoa C, Parra L, Gutierrez A, Martinez-Jimenez C, Gonzalez-Martin JM, Fernandez RL, Kacmarek RM; Stratification and Outcome of Acute Respiratory Distress Syndrome (STANDARDS) Network. Is Overall Mortality the Right Composite Endpoint in Clinical Trials of Acute Respiratory Distress Syndrome? Crit Care Med. 2018 Jun;46(6):892-899. doi: 10.1097/CCM.0000000000003022. PMID 29420341
- [Derived] Villar J, Blanco J, del Campo R, Andaluz-Ojeda D, Diaz-Dominguez FJ, Muriel A, Corcoles V, Suarez-Sipmann F, Tarancon C, Gonzalez-Higueras E, Lopez J, Blanch L, Perez-Mendez L, Fernandez RL, Kacmarek RM; Spanish Initiative for Epidemiology, Stratification & Therapies for ARDS (SIESTA) Network. Assessment of PaO(2)/FiO(2) for stratification of patients with moderate and severe acute respiratory distress syndrome. BMJ Open. 2015 Mar 27;5(3):e006812. doi: 10.1136/bmjopen-2014-006812. PMID 25818272
- [Derived] Villar J, Perez-Mendez L, Lopez J, Belda J, Blanco J, Saralegui I, Suarez-Sipmann F, Lopez J, Lubillo S, Kacmarek RM; HELP Network. An early PEEP/FIO2 trial identifies different degrees of lung injury in patients with acute respiratory distress syndrome. Am J Respir Crit Care Med. 2007 Oct 15;176(8):795-804. doi: 10.1164/rccm.200610-1534OC. Epub 2007 Jun 21. PMID 17585106